CLINICAL TRIAL: NCT04666597
Title: CariesCare International Adapted for the Pandemic in Children: Caries OUT Multicentre Single-group Interventional Study
Brief Title: Pandemic-adapted Caries Care Multicentre Single-group Interventional Study
Status: Completed | Type: Observational
Sponsor: Universidad El Bosque, Bogotá (Other)
Collaborators: King's College London (Other); University of Leeds (Other); University of Sheffield (Other)
Responsible Party: Principal Investigator, Stefania Martignon, Principal Investigator, Universidad El Bosque, Bogotá
Other Study IDs: IRB00010617
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Dental Caries in Children
Keywords: Dental caries; Children; COVID-19; Dental care; Conservative care; Aerosols; Remote consultation; Outcome assessment; Multicenter study
MeSH Terms: conditions — Dental Caries; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adapted-CCI single-intervention group in children: The single-group intervention will be the adapted-CCI 4D-cycle caries care, with non-AGP and reduced in-office appointments' time. A trained examiner per centre will conduct examinations at baseline, at 5-5.5 months (three months after basic management), 8.5 and 12 months, assessing the child's CCI caries risk and oral-health behaviour, visually staging and assessing caries-lesions severity and activity without air-drying (ICDAS-merged Epi); fillings/sealants; missing/dental-sepsis teeth, and tooth symptoms, synthetizing together with parent and external-trained dental practitioner (DP) the patient- and tooth-surface level diagnoses and personalised care plan. DP will deliver the adapted-CCI caries care. Parents' and dentists' process acceptability will be assessed via Treatment-Evaluation-Inventory questionnaires, and costs in terms of number of appointments and activities. Twenty-one centres in 13 countries will participate.
  Interventions: Procedure: Modified CariesCare International management

INTERVENTIONS:
Procedure: Modified CariesCare International management — Interventions of this single-group study correspond to the 4D, to be implemented by the external DP, when possible with remote care and only with non-AGP:
  1. D-DETERMINE risk assessing the protective and risk factors (social/medical/behavioural and clinical), using remote tools. Additionally, the description of tooth brushing behaviours and consumption of free sugars is included.
  2. D-DETECT & ASSESS: Caries staging and activity: ICDAS-merged visual criteria Caries OUT (without using compressed air, and avoiding radiographs). Clinical risk factors are assessed as well.
  3. D-DECIDE a personalized care plan: individually designed for caries management home and clinical approaches.
  4. D-DO: Appropriate Tooth-preserving & Patient-level caries: Management plan at the Patient and at the Lesion level and the implementation of the Change Behaviour Tool (CBT) designed for this protocol.
  The follow-up data will include a T1, T2 and T3 assessment.

SUMMARY:
The current understanding of dental caries has not been completely transferred into the clinical practice to control caries lesion progression (severity / activity) and the individual risk of caries. This situation led to the development of the CariesCare International CCI Caries Management System (2018), derived from ICCMS™- International Caries Classification and Management System (2012) and the ICDAS - International Caries Detection and Assessment System (2002) in a consensus among more than 45 cariologists, epidemiologists, public health professionals, researchers and cliniciansfrom all over the world. The consensus aimed to guide dentists and dental teams in clinical practice, facilitating the control of the caries process and the maintenance of oral health in their patients.

The general lack of implementation of an updated management of dental caries is evident in Colombia, in the survey of 1094 clinicians, teachers and students, failures were reported to adopt related behaviours, motivation barriers (remuneration), opportunity (in terms of relevance, physical/infrastructure resources, time) and training. As an additional barrier, the Colombian Chapter of the Alliance for a Cavity-Free Future (ACFF), evidences the absence of a facilitating Oral Health Record (OHR), this situation lead to stablish a new Alliance between the Ministry of Health and Social Protection (MSPS) and the AFLC to develop an inter-institutional consensus at the national level, of a clinical history for diagnosis and management of lesions and caries risk. Finally, 55 institutions participated in this consensus, and we have just finished a pilot test of the forms to submit a proposal for national standardization from the MSPS.

The aim of this multicentre case series is to assess after 3, 6 and 12 months in children oral health outcomes, caregivers' satisfaction and in dentists' process outcomes, after the implementation of the CCI system adapted for the COVID-19 era -non-aerosol generating procedures. Oral health outcomes will be evaluated in terms of:

* Effectiveness of CCI to control bacterial plaque, caries progression and caries risk, and to achieve behavioural change in oral health in children.
* Acceptance of CCI caries management adapted for COVID-19 through Treatment Evaluation Interventory in dentists, and in children/parents through satisfaction questionnaire.
* Costs of CCI adapted for caries management, in economic terms, number and appointment time.

DETAILED DESCRIPTION:
This study has been planned to be developed in 21 centres: 5 Colombian, 14 international dental schools, 1 Colombian health care provider and a demonstrative centre of the ACFF. Each center will implement the CCI management adapted for COVID-19 era in a total of 20 3 to 5- and 6 to 8-year-old children. Children's caries care can be delivered at dental schools' clinics and private practice. Follow-up assessments will be conducted at 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Children 3 to 5 and 6 to 8 years of age.

Exclusion Criteria:

* Family plans to move during the study time
* Oral-health related systemic conditions or physical/mental disabilities
* Presence of orthodontic/orthopaedic appliances
* Presence of MIH in first permanent molars with indication of extraction
* Children attending for a dental emergency/urgency

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants will be enrolled from the University Dental clinics, dental health providers and dental private practice across 21 multi-centre sites. The parents/caregivers of patients, aged 3 to 5 years and 6 to 8 years will be invited by the dentist to participate in the study and that their children are eligible to be considered for recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Mean number of tooth surfaces with avoidance of caries progression (ICDAS-merged Epi severity and/or activity) | up to 12 months
  With the implementation of the CCI 4D-cycle adapted for the COVID-19 pandemic characterized by the patient-centred risk -based caries management systems, the the primary outcomes consist of: At the tooth surface level in avoidance of individuals and average number of surfaces with caries progression. At the individual level consist in avoidance of caries risk level increase/no control, plaque control, and avoidance of extraction, pain, failure of the restoration. Figures will be described using mean and standard deviation (SD) for quantitative variables and percentages for qualitative variables.

SECONDARY OUTCOMES:
Proportion of subjects with avoidance of caries progression (ICDAS-merged Epi severity and/or activity) | up to 12 months
  Figures will be described using mean and standard deviation (SD) for quantitative variables and percentages for qualitative variables.
Proportion of subjects with avoidance of caries risk level increase/no control, and avoidance of extraction, pain, failure of the filling/sealant. | up to 12 months
  Figures will be described using mean and standard deviation (SD) for quantitative variables and percentages for qualitative variables.
Proportion of parents and dentists with high dental care process acceptability (measured with TEI). | up to 12 months
  Figures will be described using mean and standard deviation (SD) for quantitative variables and percentages for qualitative variables.
Proportion of subjects with avoidance of caries risk level increase/no control, and avoidance of extraction, pain, failure of the filling/sealant | up to 12 months
  Figures will be described using mean and standard deviation (SD) for quantitative variables and percentages for qualitative variables.
Proportion of children improving oral-health related behaviours | up to 12 months
  Figures will be described using mean and standard deviation (SD) for quantitative variables and percentages for qualitative variables.
Description of dental care costs | up to 12 months
  The providers' payment model of the centre will be described (Fee-for-service, Capitation, Salary-based and Pay-for-performance) (43). For the description of costs, these will be converted to the United States Dollar (USD) under the average Market Representative Exchange Rate for the year 2021 (MRER-average).

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Martignon, PhD, Principal Investigator — Universidad El Bosque
Locations (21):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - Tufts University, Boston, Massachusetts
- Argentina (2):
  - Universidad de Buenos Aires, Buenos Aires
  - Universidad Nacional de Córdoba, Córdoba
- University of Sao Paulo, São Paulo, Brazil
- Colombia (7):
  - Universidad El Bosque, Bogotá, Bogotá DC
  - Viva 1A IPS Health Provider, Barranquilla
  - Fundación Universitaria de Colegios de Colombia, Bogotá
  - Corporación Universitaria Rafael Núñez, Cartagena
  - Universidad de Cartagena, Cartagena
  - ACFF Colombian Chapter Manizales Demonstration Territory, Manizales
  - Universidad Cooperativa de Colombia, Medellín
- Universidad Iberoamericamericana, Santo Domingo, Dominican Republic
- Universite Cote d' Azur, Nice, France
- Universidad de Guadalajara, Guadalajara, Mexico
- ACTA, Amsterdam, Netherlands
- Universidad Peruana Cayetano Heredia, Lima, Peru
- University of Porto, Porto, Portugal
- University of Moscow, Moscow, Russia
- University of Sheffield, Sheffield, United Kingdom
- Universidad Católica de Uruguay, Buenos Aires, Sanmartin, Uruguay

IPD SHARING:
Plan to Share IPD: Yes
All IPD
Supporting Information: Study Protocol
Time Frame: CariesCare International adapted for the pandemic in children: Caries OUT multicentre single-group interventional study protocol

REFERENCES:
- [Result] Martignon S, Cortes A, Douglas GVA, Newton JT, Pitts NB, Avila V, Usuga-Vacca M, Gamboa LF, Deery C, Abreu-Placeres N, Bonifacio C, Braga MM, Carletto-Korber F, Castro P, P Cerezo M, Chavarria N, Cifuentes OL, Echeverri B, Jacome-Lievano S, Kuzmina I, Lara JS, Manton D, Martinez-Mier EA, Melo P, Muller-Bolla M, Ochoa E, Osorio JR, Ramos K, Sanabria AF, Sanjuan J, San-Martin M, Squassi A, Velasco AK, Villena R, Zandona AF, Beltran EO. CariesCare International adapted for the pandemic in children: Caries OUT multicentre single-group interventional study protocol. BMC Oral Health. 2021 Jul 1;21(1):329. doi: 10.1186/s12903-021-01674-1. PMID 34210281